CLINICAL TRIAL: NCT04562779
Title: Single-dose Interventions to Reduce Re-admissions for Hospitalized Patients With Refractory Alcohol Use Disorder: A Randomized Pilot Feasibility Study.
Brief Title: Inpatient Single Dose Interventions for Alcohol Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2008
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Use Disorder, Severe
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- XR Naltrexone (Experimental): Participants will receive a single dose of extended-release, injectable naltrexone prior to hospital discharge, in addition to enhanced linkage to follow-up addiction care.
  Interventions: Drug: Naltrexone 380 MG; Behavioral: Enhanced linkage
- IV Ketamine (Experimental): Participants will receive a single dose of intravenous ketamine (0.5mg/kg over 40 minutes) prior to hospital discharge, in addition to enhanced linkage to follow-up addiction care.
  Interventions: Drug: Ketamine Hydrochloride; Behavioral: Enhanced linkage
- Linkage (Active Comparator): Participants will receive no single-dose addiction medication prior to hospital discharge, but will receive enhanced linkage to follow-up addiction care.
  Interventions: Behavioral: Enhanced linkage

INTERVENTIONS:
Drug: Naltrexone 380 MG — XR naltrexone to be given once prior to hospital discharge
  Arms: XR Naltrexone
Drug: Ketamine Hydrochloride — IV ketamine infusion to be given once prior to hospital discharge
  Arms: IV Ketamine
Behavioral: Enhanced linkage — Includes in-hospital intake at outpatient addiction clinic plus contingency management related to follow-up

SUMMARY:
Every year, alcohol use disorder (AUD) generates millions of emergency department (ED) visits and hospital admissions, costing the U.S. health sector over $90 billion. These hospital admissions are critical opportunities to start patients on addiction pharmacotherapy, but factors like medication non-adherence and post-discharge relapse contribute to frequent re-admissions. Two single-dose interventions are well suited to facilitate treatment retention and prevent re-admissions due to their prolonged, adherence-independent effects: extended-release (XR) naltrexone injection and intravenous (IV) ketamine infusion. These have not been thoroughly investigated in the hospital setting among high-utilizer, safety-net populations. Therefore, the investigators aim to:

1. Test the feasibility of randomizing hospitalized patients (n=45-60, age 18-65) with multiple AUD-related admissions to treatment with either extended-release (XR) naltrexone, intravenous (IV) ketamine, or no single-dose medication, all with enhanced linkage to care. Feasibility outcomes such as recruitment rate, patient acceptability, post-discharge follow-up rate, and adverse events will help to identify key lessons for a future comparative effectiveness study.
2. Estimate the 30-day re-admission rate for patients randomized to treatment with XR naltrexone, with IV ketamine, or no single-dose medication, all with enhanced linkage to care. The investigators hypothesize that the re-admission rate will be lower for each of the two single-dose medication groups than for the "linkage-alone" group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* 1+ alcohol-related* admission(s) or emergency department visit(s) in past 12 mo.
* Has insurance (public or private)
* Seen by inpatient addiction consult service

Exclusion Criteria:

* Known or suspected active COVID-19 infection
* Hepatic: AST/ALT >5x upper-limit of normal, decompensated liver failure
* Renal: Glomerular filtration rate <30ml/min
* Cardiovascular: History of acute coronary syndrome, cerebrovascular event, hypertensive crisis, known cardiomyopathy
* Known elevated intracranial pressure
* Thrombocytopenia (<50/microliter)
* Active moderate/severe withdrawal (based on hospital withdrawal protocol)
* Active delirium (alcohol-related or otherwise)
* Already enrolled in study
* XR naltrexone or IV ketamine in last 30 days
* Known intolerance to naltrexone or ketamine
* Other active severe substance use disorder (tobacco, cannabis excluded)
* Pregnant or breast-feeding, or planning.
* Opioids: chronic, recent (<24h), or anticipated
* Unstable psychiatric illness (active psychosis, active suicidality)
* Moving from region within 30-days of discharge
* Discharge to acute/residential treatment
* Involuntary hold

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terasaki D, Loh R, Cornell A, Taub J, Thurstone C. Single-dose intravenous ketamine or intramuscular naltrexone for high-utilization inpatients with alcohol use disorder: pilot trial feasibility and readmission rates. Addict Sci Clin Pract. 2022 Nov 22;17(1):64. doi: 10.1186/s13722-022-00345-y. PMID 36419181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital.
Period: Overall Study
Arm/Group | XR Naltrexone | IV Ketamine | Linkage
Started | 14 | 13 | 17
Completed | 5 | 6 | 7
Not Completed | 9 | 7 | 10
Not completed — Lost to Follow-up | 7 | 5 | 10
Not completed — Protocol Violation | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XR Naltrexone | IV Ketamine | Linkage | Total
Number analyzed (Participants) | 14 | 13 | 17 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.5) | 43.9 (11.5) | 46.2 (9.5) | 45.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 11 | 9 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 5 | 15
  Not Hispanic or Latino | 8 | 8 | 12 | 28
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 2 | 7
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 4 | 9 | 12 | 25
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 4 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 17 | 44

OUTCOME MEASURES:

1. Primary Outcome: Rate (%) of 30-day Hospital Re-admission
Description: Binary outcome: any all-cause hospitalization ascertained by chart review (our EHR includes records from several local hospitals).
  Note that it is not dependent on study completion, so it is analyzed by intent to treat.
Time Frame: Within 30 days of index hospital discharge. The enrollment period is 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | XR Naltrexone | IV Ketamine | Linkage
Number analyzed (Participants) | 14 | 13 | 17
Participants | 3 | 2 | 7

2. Primary Outcome: Feasibility - Recruitment Rate (# Per Month)
Description: Number of participants recruited per month during the enrollment period
Time Frame: The enrollment period is 12 months
Measure: Mean (Standard Deviation); unit: participants per month recruited
Groups:
- Full Trial Sample: Full trial sample
Arm/Group | Full Trial Sample
Number analyzed (Participants) | 44
participants per month recruited | 3.7 (2.8)

3. Primary Outcome: Feasibility - Follow-up Rate (%)
Description: Percentage of patients who presented to follow-up appointment within 14 days
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | XR Naltrexone | IV Ketamine | Linkage
Number analyzed (Participants) | 14 | 13 | 17
Participants | 7 | 8 | 7

4. Secondary Outcome: Rate (%) of 30-day Emergency Department Visit
Description: Binary outcome: any all-cause ED visit ascertained by chart review
Time Frame: Within 30 days of index hospital discharge. The enrollment period is 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | XR Naltrexone | IV Ketamine | Linkage
Number analyzed (Participants) | 14 | 13 | 17
Participants | 8 | 7 | 12

ADVERSE EVENTS:
Time Frame: Immediate effects of IM naltrexone or IV ketamine were assessed immediately after administration in the hospital. Adverse events by PRISE questionnaire were assessed at follow-up visit (targeted at 1 week post-discharge) for those who attended. Deaths and serious adverse events would be detected at any point within 30 days post-discharge from electronic health record alerts, direct patient communication with study team, or other staff communication.
Description: Hospital admission or emergency department visits were not automatically considered serious adverse events. This is because these were the primary/secondary outcomes targeted by the intervention itself.
Arm/Group | XR Naltrexone | IV Ketamine | Linkage
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 5/14 | 6/13 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XR Naltrexone (N=14) | IV Ketamine (N=13) | Linkage (N=17)
diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 — tolerable
diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 — distressing
constipation (Gastrointestinal disorders) | 1 | 2 | 0 — tolerable
constipation (Gastrointestinal disorders) | 0 | 0 | 0 — distressing
dry mouth (Gastrointestinal disorders) | 1 | 2 | 2 — tolerable
dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 — distressing
nausea/vomiting (Gastrointestinal disorders) | 1 | 1 | 1 — tolerable
nausea/vomiting (Gastrointestinal disorders) | 1 | 0 | 0 — distressing
abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 — tolerable
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 — distressing
increased appetite (Gastrointestinal disorders) | 3 | 3 | 2 — tolerable
decreased appetite (Gastrointestinal disorders) | 4 | 0 | 0 — tolerable
decreased appetite (Gastrointestinal disorders) | 0 | 0 | 1 — distressing
palpitations (Cardiac disorders) | 1 | 1 | 1 — tolerable
palpitations (Cardiac disorders) | 1 | 0 | 0 — distressing
dizziness on standing (Cardiac disorders) | 2 | 3 | 3 — tolerable
dizziness on standing (Cardiac disorders) | 1 | 0 | 0 — distressing
chest pain (Cardiac disorders) | 2 | 1 | 0 — tolerable
chest pain (Cardiac disorders) | 1 | 0 | 0 — distressing
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — tolerable
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 — distressing
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 — tolerable
cough (Reproductive system and breast disorders) | 0 | 0 | 1 — distressing
pain with breathing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 — tolerable
pain with breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 — distressing
injection site reaction (naltrexone) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — tolerable
injection site reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — distressing
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — tolerable
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — distressing
increased perspiration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — tolerable
increased perspiration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — distressing
itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 — tolerable
itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — distressing
dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 — tolerable
dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — distressing
headache (Nervous system disorders) | 2 | 1 | 1 — tolerable
headache (Nervous system disorders) | 1 | 0 | 0 — distressing
tremor (Nervous system disorders) | 0 | 0 | 2 — tolerable
tremor (Nervous system disorders) | 1 | 1 | 2 — distressing
poor coordination (Nervous system disorders) | 2 | 3 | 3 — tolerable
poor coordination (Nervous system disorders) | 1 | 0 | 0 — distressing
dizziness or lightheadedness (Nervous system disorders) | 3 | 2 | 2 — tolerable
dizziness or lightheadedness (Nervous system disorders) | 0 | 0 | 0 — distressing
numbness or tingling (Nervous system disorders) | 2 | 1 | 2 — tolerable
numbness or tingling (Nervous system disorders) | 0 | 0 | 0 — distressing
speech difficulty (Nervous system disorders) | 2 | 0 | 0 — tolerable
speech difficulty (Nervous system disorders) | 1 | 0 | 0 — distressing
blurred vision (Eye disorders) | 1 | 2 | 2 — tolerable
blurred vision (Eye disorders) | 1 | 0 | 2 — distressing
ringing in ear (Ear and labyrinth disorders) | 0 | 1 | 1 — tolerable
ringing in ear (Ear and labyrinth disorders) | 0 | 0 | 0 — distressing
difficulty urinating (Renal and urinary disorders) | 0 | 0 | 2 — tolerable
difficulty urinating (Renal and urinary disorders) | 0 | 0 | 0 — distressing
painful urination (Renal and urinary disorders) | 0 | 0 | 0 — tolerable
painful urination (Renal and urinary disorders) | 0 | 0 | 0 — distressing
frequent urination (Renal and urinary disorders) | 1 | 3 | 3 — tolerable
frequent urination (Renal and urinary disorders) | 0 | 0 | 0 — distressing
menstrual irregularity (Reproductive system and breast disorders) | 0 | 0 | 0 — tolerable
menstrual irregularity (Reproductive system and breast disorders) | 0 | 0 | 0 — distressing
increased libido (Reproductive system and breast disorders) | 0 | 2 | 0 — tolerable
increased libido (Reproductive system and breast disorders) | 0 | 0 | 0 — distressing
decreased libido (Reproductive system and breast disorders) | 1 | 1 | 1 — tolerable
decreased libido (Reproductive system and breast disorders) | 0 | 1 | 0 — distressing
difficulty sleeping (Psychiatric disorders) | 2 | 3 | 3 — tolerable
difficulty sleeping (Psychiatric disorders) | 1 | 1 | 0 — distressing
abnormal dreams (Psychiatric disorders) | 3 | 4 | 1 — tolerable
abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 — distressing
anxiety (Psychiatric disorders) | 2 | 3 | 4 — tolerable
anxiety (Psychiatric disorders) | 4 | 2 | 1 — distressing
hallucinations (Psychiatric disorders) | 1 | 1 | 1 — tolerable
hallucinations (Psychiatric disorders) | 0 | 0 | 1 — distressing
memory loss (Psychiatric disorders) | 2 | 2 | 0 — tolerable
memory loss (Psychiatric disorders) | 1 | 1 | 1 — distressing
poor concentration (Psychiatric disorders) | 3 | 1 | 3 — tolerable
poor concentration (Psychiatric disorders) | 1 | 2 | 0 — distressing
fatigue or decreased energy (General disorders) | 4 | 0 | 3 — tolerable
fatigue or decreased energy (Psychiatric disorders) | 1 | 2 | 0 — distressing
restlessness (General disorders) | 4 | 2 | 0 — tolerable
restlessness (General disorders) | 1 | 2 | 0 — distressing
other (General disorders) | 1 | 0 | 0 — tolerable
other (General disorders) | 0 | 0 | 0 — distressing
increased appetite (Gastrointestinal disorders) | 0 | 0 | 0 — distressing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04562779/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04562779/ICF_001.pdf